CLINICAL TRIAL: NCT04618003
Title: Analysis of Autonomic Modulation in Athletes and Non-Athletes With Spinal Cord Injury During Task in Virtual Reality Environment
Brief Title: Autonomic Modulation in Athletes and Non-Athletes With Spinal Cord Injury During Task in Virtual Reality Environment
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Talita Dias da Silva, Researcher, University of Sao Paulo
Other Study IDs: 79346017.8.0000.5505
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Athletes with Spinal Cord Injury: Group of athletes with spinal cord injury that was assessed at rest and during a physical activity in virtual reality.
  Interventions: Behavioral: Adaptation of autonomic nervous system to activity in virtual reality
- Non-athletes with spinal cord injury: Group of non-athletes with spinal cord injury that was assessed at rest and during a physical activity in virtual reality.
  Interventions: Behavioral: Adaptation of autonomic nervous system to activity in virtual reality
- Able-bodied control group: Group of non-athletes able-bodied control subjects that was assessed at rest and during a physical activity in virtual reality.
  Interventions: Behavioral: Adaptation of autonomic nervous system to activity in virtual reality

INTERVENTIONS:
Behavioral: Adaptation of autonomic nervous system to activity in virtual reality — heart rate variability assessed at rest and during a physical activity in virtual reality.

SUMMARY:
The study consisted in the analysis of the autonomic modulation of the heart rate by the Heart Rate Variability of the participants at rest for 5 minutes, and during physical activity of 8 minutes, through a virtual reality game. The data capture was performed using a cardio-frequency meter with belt placed on the volunteer's trunk and, in addition, questionnaires, functional classification scales and personal data collection were applied.

DETAILED DESCRIPTION:
This is a cross-sectional study, approved by the Ethics and Research Committee of the Medical School of the Federal University of São Paulo (UNIFESP) registered under CAAE 793517.1.0000.5505. The recruitment of non-athletes was carried out at the Acreditando Rehabilitation Center and the athletes were recruited at the Faca na Cadeira Institute, ICEL and Clube Espéria. Participants were enrolled in the study after signing the Free and Informed Consent Term. Convenience sampling technique was used with data collected from March 2017 to October 2018 Participants The study included athletes and non-athletes with a confirmed medical diagnosis of SCI, with voluntary extension of elbows and wrist, active trunk control, and who had already completed rehabilitation. For the athlete group, participants had to fulfill the minimum criteria for defining an active athlete, described in the next section. Also, a control group of able-bodied subjects, approximately paired by age and sex wit the AG and non-athlete groups were recruited. Participants were excluded if they presented with impairments to the upper limbs that interfered with the performance during the game, were diagnosed with heart disease or other neurological disorders , were using medication that were not part of their usual routine or that influenced the cardiac and nervous systems, and presented an error greater than 5% in the analysis of HRV.

Assessment of function The Funtional Independence Measure (FIM) and the Spinal Cord Independence Measure Version III (SCIM III) were used to classify functional independence. The International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) was employed to assess the level and severity of injury. To classify the physical activity levels of the participants, the the Physical Activity in Athlete Questionnaire and the Leisure Time Physical Activity Questionnaire for Non-Athletes with Spinal Cord Injury (LTPAQ-SCI) were employed.

Assessment of Heart Rate Variability For the HRV assessment, participants were instructed not to consume alcohol, caffeine or smoke 24 hours before the test. The procedures to measure HRV were conducted according to the guidelines from the Task Force of the European Society of Cardiology and the North American Society of Stimulation and Electrophysiology and were recorded using the Polar V800 electrocardiographic measuring device (Polar Electro, Finland), with a sampling rate of 1000 Hz.

The determination of the linear indexes of HRV for time and frequency was carried out using the software Kubios HRV (v. 3.3.0). The HRV data for time was analyzed using linear methods, using SDNN indices (standard deviation of the mean of all normal RR intervals) in milliseconds (ms); PNN50 (percentage of successive differences of the RR intervals with an absolute value greater than 50ms); RMSSD (square root of the mean square of the differences between adjacent normal RR intervals). Moreover, geometric methods such as, the RRTri (triangular index) and TINN (histogram interpolation of NN intervals), the indexes of the Poincaré graph with the SD1 (standard deviation of the instantaneous variability of the beat-to beat heart rate), SD2 (standard deviation of the long-term, continuous, RR interval variability), and the SD1/SD2 ratio-the ratio between the short- and long-term variations among the RR intervals and Parassympathetic Nervous System index (PNS index), Sympathetic Nervous System index (SNS index) and Stress index given by HRV Kubios, were employed. LF indices (low frequency spectral components, between 0.04 and 0.15 Hertz) were recorded in ms2 and in standard units (nu); while HF (high frequency spectral components, between 0.15 and 0.4 Hertz) was recorded in ms2 and nu; and the ratio of LF/HF in ms2.

PROTOCOL For the three groups the HRV measures were captured in 2 instances: 1. For 5 minutes at rest in the seated position; and 2. During the VR activity, in which the individual executed movements according to a game in front of a computer for 8 minutes. The VR activity was performed using the game MoveHero, developed at the School of Arts Sciences and Humanities of the University of São Paulo (EACH-USP). The game consists of virtual balls that fall in pre-determined time intervals and spacial distribution in four imaginary columns on a computer screen. The participant must move in the direction of the balls to touch them as they reach four pre-determined targets placed to the sides of the player's avatar. The targets are numbered (1 to 4) and are placed in parallel at two different heights, two to the left and two to the right of the player's avatar.

The game captures the participant's movements with a webcam, not requiring physical contact to perform the task. The participant must move his arms at 80% of their maximum lateral range. Before starting the task, the experimenter positioned the participant in a distance from the screen that allowed him/her to achieve the maximum lateral reach range for each side (left and right) when reaching towards the two farthest balls (1 and 4). From that position, the distance between the computer's table and the participant's feet was measured and the participant was asked to move his/her wheelchair to 80% of this distance. During the task, the participant had to wait for the balls to drop until they reached the pre-determined targets. When the balls reached the targets, the color of the balls changed to green, which prompted the participant to reach for them. Therefore, the game requires the participant to have a strategy of planning their movement to reach the targets at the same time as the balls.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed medical diagnosis of SCI
* Preserved motor activity for extension of the upper limbs and active trunk control, which had already finished their process of adaptation to injury.

Exclusion Criteria:

* Functional incapacities of the upper limbs to perform the game,
* Diagnosis of heart disease or other neurological disorders not due to SCI,
* Consumption of drugs that are not part of their usual treatment routine and that influence the cardiac and nervous systems,
* Error greater than 5% in the analysis of HRV.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study included athletes and non-athletes with a confirmed medical diagnosis of SCI, with voluntary extension of elbows and wrist, active trunk control, and who had already completed rehabilitation. For the athlete group, participants had to fulfill the minimum criteria for defining an active athlete, described in the next section. Also, a control group of able-bodied subjects, approximately paired by age and sex wit the and non-athlete groups were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Cardiac autonomic modulation is different between athletes and non athletes with spinal cord injury (SCI), bu no differences between athletes with SCI and able-bodied controls. | 1 day
  Athletes with SCI present a better cardiac autonomic modulation then non-athletes with SCI, assessed through linear and non-linear heart rate variability indices at rest and during VR activity
Athletes and able-bodied subjects present a good adaptation of autonomic nervous system than non-athletes with spinal cord injury. | 1 day
  Athletes and able-bodied controls present a good adaptation of autonomic nervous system assessed through indices of heart rate variability. i.e. parasympathetic withdraw during physical activity in Virtual Reality, but with no significant difference for non-athletes with spinal cord injury.

CONTACTS AND LOCATIONS:
Overall Officials: Talita D Silva, Ph.D., Principal Investigator — University of Sao Paulo
Locations (1):
- Comitê de Ética e Pesquisa da Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dias ED, de Menezes LDC, da Silva TD, da Silva NM, Vidal PR, Brondane BR, Padula N, Gaspar RC, Santos S, Auricchio JR, de Mello Monteiro CB, Domingo A, de Oliveira CQ, de Macedo JC, Romanholo BMS, Barnabe V. Comparison of cardiac autonomic modulation of athletes and non-athletes individuals with spinal cord injury at rest and during a non-immersive virtual reality task. Spinal Cord. 2021 Dec;59(12):1294-1300. doi: 10.1038/s41393-021-00722-5. Epub 2021 Nov 2. PMID 34728783